CLINICAL TRIAL: NCT01876186
Title: Comparisons of Urodynamic Effects, Urinary Nerve Growth Factor Levels and Outcomes in Female Overactive Bladder Patients After 3-month Versus 6-month Solifenacin Treatment: a Randomized Prospective Study
Brief Title: Comparisons of 3-month Versus 6-month Solifenacin Treatment for Female OAB Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201212143RINB
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Overactive Bladder Syndrome
Keywords: antimuscarinic treatment; urodynamic studies; nerve growth factor
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solifenacin for 12 weeks group (Experimental): Solifenacin (5 mg qd) for 12 weeks
  Interventions: Drug: Solifenacin for 12 weeks
- Solifenacin for 24 weeks group (Active Comparator): Solifenacin (5 mg qd) for 24 weeks
  Interventions: Drug: Solifenacin for 24 weeks

INTERVENTIONS:
Drug: Solifenacin for 12 weeks — Solifenacin 5 mg one a day for 12 weeks
  Other Names: Vesicare
  Arms: Solifenacin for 12 weeks group
Drug: Solifenacin for 24 weeks — Solifenacin 5 mg once a day for 24 weeks
  Other Names: Vesicare
  Arms: Solifenacin for 24 weeks group

SUMMARY:
To investigate whether prolonged period of treatment (6 months) can have a better therapeutic outcome than conventional period (3 months) of antimuscarinics.

DETAILED DESCRIPTION:
Overactive bladder syndrome (OAB), with or without urge incontinence, is characterized by urinary urgency, frequency and nocturia. Thus, patients with OAB could be considered to have a reduced quality of life. Patients with overactive bladder syndrome have a higher risk of falling and fracture due to nocturia. OAB affects around 17 % of female population. At present, muscarinic receptor antagonists are the ﬁrst-line pharmacotherapeutic agents for OAB. However, discontinuation of the treatment often results in symptom relapse. Until now, optimal duration of the treatment and durability of the efﬁcacy have not been determined. We plan to use urodynamic studies outcome to evaluate therapeutic effect, with the change of urinary nerve growth factor level. This study is a randomized prospective study, comparing female OAB patient after 3 months and 6 months of antimuscarinic treatment.

The purpose of this study is to investigate the difference of urodynamic effects, therapeutic effect and urinary urinary nerve growth factor level between OAB females after 3 months and 6 months antimuscarinic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women who have overactive bladder syndrome

Exclusion Criteria:

* Women who are less than 20 year-old

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The rate of normalized urodynamic findings | 6 months
  The rate of normalized urodynamic finding after antimuscarinics

SECONDARY OUTCOMES:
The cure rate of overactive bladder | 24 weeks
  The cure rate of overactive bladder after antimuscarinics
The recurrence rate of overactive bladder | 2.5 years
  The recurrence rate of overactive bladder after antimuscarinics
The difference of urine nerve growth factor level | 24 weeks
  The difference of urine nerve growth factor level after antimuscarinics

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan